CLINICAL TRIAL: NCT06152796
Title: Paracetamol Versus Ibuprofen in Closure of Patent Ductus Arteriosus in Premature Neonates,at Upper Egypt
Brief Title: Comparision Between Paracetamol and Ibuprofen in Closure of Patent Ductus Arteriosus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Abdelfatah Abdelaal Abdelsamie, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: closure of PDA
Record Dates: First submitted 2023-11-15; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol (Experimental): preterms receive oral/iv paracetamol at the dose of 15 mg/kg every 6 h for 3 days.
  Interventions: Drug: Paracetamol
- Ibuprofen (Experimental): preterms receive oral ibuprofen at the initial dose 10 mg/kg, followed by 5 mg/kg after 24 and 48 h
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Paracetamol — Anti_inflammatory drug
  Arms: Paracetamol
Drug: Ibuprofen — Non steroidal anti_inflammatory drug
  Arms: Ibuprofen

SUMMARY:
To compare efficacy and safety of paracetamol and ibuprofen for the pharmacological closure of patent ductus arteriosus (PDA) in preterm infants.

DETAILED DESCRIPTION:
The ductus arteriosus (DA) is an essential fetal blood vessel that connects the pulmonary artery to the aorta and serves to shunt blood away from the lungs into the umbilical placental circulation where gas exchange takes place.At birth, closure of the DA is a critical event in the transition to the postnatal circulatory pattern. However, there are situations in which DA closure does not occur or is delayed, resulting in the condition known as persistent patent DA (PDA) .

After birth, it usually closes within 48 h. A persistently PDA is diagnosed when the DA fails to close after 72 h.

PDA accounts for 5% to 10% of all congenital heart diseases. However, the incidence surges up to 60% in preterm infants and is inversely related to gestational age(GA) and birth weight.

The closure of the DA in full-term infants occurs in two steps. Initially, within the first few hours after birth,increased arterial PaO2 and decreased circulating prostaglandins allow the smooth muscle media of the ductus to constrict. As a result of the constriction, the inner muscle wall of the DA develops profound ischemic hypoxia which leads to the formation of vascular endothelial growth factor, transforming growth factor beta,and other inflammatory mediators and growth factors that transform the ductus into a non-contractile ligament.

The clinical consequences of PDA are related to the degree of left- to-right shunting through the PDA, with its associated change in blood flow to the lungs, kidneys, and intestine . This results in increased pulmonary blood flow and increased incidence of further comorbidities such as chronic lung disease, intraventricular hemorrhage(IVH), necrotizing enterocolitis (NEC), and retinopathy.Therefore, closure of the PDA is essential to prevent these complications and to improve both cardiorespiratory status and survival rate .

Clinical criteria of hemodynamically significant PDA (hs-PDA) are the following: tachycardia,bounding pulse with wide pulse pressure, hyperdynamic precordium with continuous murmur on auscultation, hepatomegaly, edema, unexplained metabolic acidosis, failure of respiratory distress syndrome to improve at 2-7 days, and unexplained CO2 retention in mechanically ventilated neonates.

Echocardiography has been examined in multiple studies as an objective measure of hs-PDA.Echocardiographic criteria of hs-PDA are the following: left atrial dilatation (left atrial: aortic root >1.6), diastolic turbulence (backflow) on Doppler in the pulmonary artery, internal diameter of duct >1.5 mm, and reverse end diastolic flow in the descending aorta/mesenteric artery .

Treatment options for hs-PDA include conservative management, pharmacologic interventions, surgical ligation, and a transcatheter approach to ductal closure. However, a consensus on PDA management strategies remains elusive. Surgical ligation is usually considered when other medical treatments have either failed or were contraindicated.

For this purpose, the first-line therapy is medical and nonsteroidal anti-inflammatory drugs (NSAIDs) are drugs of choice, preventing the conversion of arachidonic acid into prostaglandins via cyclooxygenase (COX) inhibition, in both the existing isoforms COX-1 (constitutive) and COX-2 (inducible) . Reduction in prostaglandin levels leads to DA muscular wall constriction through the hypoxia of ductal vasa vasorum and consequent local angiogenesis, formation of neointimal tissue, and apoptosis. These mechanisms, in conjunction with platelet recruitment and activation, lead to processes of obstruction and fibrosis and, as a result, anatomical ductal closure .

Ibuprofen, a non-steroidal anti-inflammatory drug, inhibits both cyclooxygenase-1 and cyclooxygenase-2, which are enzymes necessary for the conversion of arachidonic acid to various prostaglandins among them PGE2.Unlike ibuprofen, paracetamol is thought to act on prostaglandin synthase at the peroxidase region of the enzyme.The role of paracetamol as an alternative treatment for the closure of hsPDA has gained attention because of the potential side-effects of cyclooxygenase inhibitors.

Studies comparing oral paracetamol versus oral ibuprofen in PDA closure reported that oral paracetamol and ibuprofen were similarly effective for the closure of PDA.While,El-Farrash et al. demonstrated that oral paracetamol is an effective and well-tolerated, first line drug treatment of PDA that was comparable to ibuprofen in terms of the rate of ductal closure and even showed decreased LPA, RVSP and LA/Ao ratio.Also,Al-Shaibi et al. documented that oral paracetamol was between cost-effective and dominant over both oral and IV ibuprofen formulations.However, another study done by Roofthooft et al.showed disappointing results with IV paracetamol administration, as PDA closure was reported in only 18% of the patients with relatively low gestational age.

Regarding the drug safety profile,Oncel et al.and Dang et al.reported that both drugs were tolerated and deemed safe in terms of renal and liver variables, as well as a lack of statistically significant difference in major complications(NEC,IVH,bronchopulmonary dysplasia).However,Balachander et al. Revealed Incidence of AKI is significantly lower with paracetamol as compared to ibuprofen.Also, Hammerman et al. reported that paracetamol could offer important therapeutic advantages over NSAIDs (e.g., indomethacin and ibuprofen), as paracetamol has no peripheral vasoconstrictive effect and can be given to infants with clinical contraindications to NSAIDs.

The availability of different management options poses a challenge for neonatologists when making evidence-based management decisions after diagnosing hemodynamically significant PDAs. The dilemma is whether to use pharmacotherapy at all, and if a decision is made to treat the PDA medically, what should be the ideal choice of pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants
* with gestational age ≤37weeks
* who had echocardiographically confirmed significant PDA.

Exclusion Criteria:

* Preterm neonates
* with major congenital anomalies,
* life threatening sepsis,
* NEC,
* IVH,
* urine output <1ml/kg/h in the last 24 h,
* serum creatinine concentration >1.5 mg/dl, -platelet count <100,000/ml,
* complex congenital heart,
* or duct-dependent lesions.

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Closure of PDA | 6 days
  Echo confirmed closure